CLINICAL TRIAL: NCT05229848
Title: Prospective Comparison of ICE Based Atrial Flutter Ablation Vs Conventional Fluoroscopy/Anatomical Mapping Based Ablation
Brief Title: ICE Based Atrial Flutter Ablation Vs Conventional Fluoroscopy/Anatomical Mapping Based Ablation - ICE Flutter Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCHRF-ICE Flutter-0010
Record Dates: First submitted 2021-12-28; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-12

CONDITIONS: Atrial Flutter
Keywords: Atrial Flutter; Ablation; Intra-cardiac echocardiogram (ICE)
MeSH Terms: conditions — Atrial Flutter | interventions — Ice

STUDY DESIGN:
Intervention Model Description: Total 60 patients will be studied. St.Jude View Flex ICE catheter and Siemens AcuNav ICE catheter are used routinely for all left sided ablation procedures which require transeptal puncture. ICE imaging catheter is typically introduced through an 11-F hemostatic sheath and positioned under fluoroscopic guidance in right atrium. After catheter coupling to the imaging platform, imaging frequency is optimized using adjunctive gain, depth, and focal length controls to define anatomic structures and minimize noise.Imaging is performed at different levels in right atrium, if needed. Imaging targets included right atrium, coronary sinus orifice, fossa ovalis, interatrial septum(IAS), tricuspid valve,left atrium, left atrial appendage, orifice of all pulmonary veins,mitral valve, papillary muscles, aortic and pulmonary valve leaflets, right ventricle, right ventricular outflow tract(RVOT),pericardial space,esophagus,aorta and adjoining left ventricular and right ventricular myocardium.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D electroanatomical mapping alone (Active Comparator): Patients who are diagnosed with typical right sided flutter who are scheduled for an ablation procedure will be enrolled. Informed consent will be obtained from each of them prior to the procedure. Patients will be randomly assigned to undergo either 3D electroanatomical mapping alone vs ICE plus 3D electroanatomical mapping guided CTI ablation. Operators will plan to alternate each case with the use of ICE + 3D mapping and 3D mapping alone with one method followed by the other for randomization. All patients will have the standard access sheaths placed in the right femoral vein.
  Interventions: Procedure: 3D electroanatomical mapping alone guided CTI ablation
- ICE plus 3D electroanatomical mapping (Experimental): Patients who are diagnosed with typical right sided flutter who are scheduled for an ablation procedure will be enrolled. Informed consent will be obtained from each of them prior to the procedure. Patients will be randomly assigned to undergo either 3D electroanatomical mapping alone vs ICE plus 3D electroanatomical mapping guided CTI ablation. Operators will plan to alternate each case with the use of ICE + 3D mapping and 3D mapping alone with one method followed by the other for randomization. All patients will have the standard access sheaths placed in the right femoral vein. The group randomized to ICE catheter placement will have a left femoral 11F sheath placed in addition.
  Interventions: Procedure: ICE plus 3D electroanatomical mapping guided CTI ablation

INTERVENTIONS:
Procedure: 3D electroanatomical mapping alone guided CTI ablation — 3D electroanatomical mapping in combination with fluoroscopy has been traditionally used in conventional CTI ablation for AFL.
  Arms: 3D electroanatomical mapping alone
Procedure: ICE plus 3D electroanatomical mapping guided CTI ablation — ICE imaging catheter is typically introduced through an 11-F hemostatic sheath and positioned under fluoroscopic guidance in the right atrium. After catheter coupling to the imaging platform, imaging frequency is optimized by the operator using adjunctive gain, depth, and focal length controls to define anatomic structures and minimize noise. Imaging is performed at different levels in the right atrium, if needed. Imaging targets included the right atrium, coronary sinus orifice, fossa ovalis, interatrial septum (IAS), tricuspid valve, left atrium, left atrial appendage, orifice of all pulmonary veins, mitral valve, papillary muscles, aortic and pulmonary valve leaflets, right ventricle, RVOT, pericardial space, esophagus, aorta and adjoining left ventricular and right ventricular myocardium.
  Arms: ICE plus 3D electroanatomical mapping

SUMMARY:
Intracardiac echocardiography (ICE), has been an essential component of Radiofrequency (RF) ablations for AF given its association with decreased fluoroscopy time and complication rates, and therefore it is logical that this can be applied to CTI ablations for AFL as well. There are however no studies to date that directly focused on the benefits of adding ICE during CTI dependent AFL ablation. Currently it is not required that operators use ICE in every case of AFL ablation. Investigators intended to study the routine use of ICE in such cases and to see if there is a significant benefit in routine use of ICE.

DETAILED DESCRIPTION:
Atrial flutter (AFL) is a re-entrant tachyarrhythmia that involves the atria that leads to both rapid ventricular rates as well as a loss of effective contractility of the atrial making them vulnerable to formation of thrombi similar to atrial fibrillation (AF). Incidence rates ranges between 5/100,000 in those <50 years old to 587/100,000 in subjects older than 80. AFL often coexists or precedes AF. In a longitudinal study, 56% of patients with lone AFL eventually developed AF. A variety of atrial flutters have been described apart from the classic cavotricuspid isthmus (CTI) dependent flutters. These include left atrial flutters and scar based reentry flutters. Atrial flutter is often a persistent rhythm that requires electrical cardioversion or radiofrequency catheter ablation for termination. While AFL may recur after cardioversion with or without antiarrhythmic therapy, ablation offers a more curative approach for this rather intolerant arrhythmia.

3D electroanatomical mapping in combination with fluoroscopy has been traditionally used in conventional CTI ablation for AFL. However, there are instances when ablation of the CTI is challenging as a result of various factors including a thick Eustachian ridge, presence of a sub-Eustachian pouch, or prominent pectinate muscles. Isthmus anatomy has been shown to affect the parameters of ablation procedure. 3D mapping to overcome difficult anatomy may not be the answer for difficult situations as shown by some operators . These anatomical challenges can not only lengthen procedural times but also lead to increased risk of complications such as perforation, effusion, or cardiac tamponade. Intracardiac echocardiography (ICE), has been an essential component of Radiofrequency (RF) ablations for AF given its association with decreased fluoroscopy time and complication rates, and therefore it is logical that this can be applied to CTI ablations for AFL as well. There are however no studies to date that directly focused on the benefits of adding ICE during CTI dependent AFL ablation. Currently it is not required that operators use ICE in every case of AFL ablation. Investigators intend to study the routine use of ICE in such cases and to see if there is a significant benefit in routine use of ICE.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing typical CTI dependent AFL who give informed consent for participation in the study will be included.

Exclusion criteria:

* Patients in whom placement of an ICE catheter in the right atrium for adequate atrial visualization is technically not feasible.
* Patients who cannot give an informed consent will be excluded.
* Patients in who vascular access for the 11F sheath is not feasible will be excluded. Those with left iliac vein stenosis or left groin arteriovenous (AV) fistulas or prior left groin access complications will be excluded.
* Patients who on the EP (Electrophysiology) study are found to have a left sided arrhythmia needing transseptal access will be excluded.
* Patients who during EP study are found to have atypical flutter pathways including Left Atrial (LA)/Left sided flutter as above, atypical pathways outside of the CTI, and scar based- reentry pathways.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Procedural duration, fluoroscopy time, and RF time assessment | These are all intraprocedural characteristics
  To assess the procedural duration, fluoroscopy time, and RF time of patients undergoing CTI dependent flutter ablation using ICE catheter along with 3D anatomical plus fluoroscopy imaging guidance compared to the same parameters in patients undergoing CTI dependent flutter ablation using only 3D anatomical plus fluoroscopy imaging guidance alone.
Post procedural complications | Post-operative Day#0-7
  To assess the incidence of post procedural complications such as incidence of perforation, pericardial effusion, cardiac tamponade, and pericarditis.
Procedural success - Number of patients with bidirectional block (entrance block and exit block) at the end of the procedure. | End of procedure marker of success
  To assess the procedural success of ablation procedures in terms of achieving bidirectional block.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (3):
- United States (3):
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Granada J, Uribe W, Chyou PH, Maassen K, Vierkant R, Smith PN, Hayes J, Eaker E, Vidaillet H. Incidence and predictors of atrial flutter in the general population. J Am Coll Cardiol. 2000 Dec;36(7):2242-6. doi: 10.1016/s0735-1097(00)00982-7. PMID 11127467
- [Background] Halligan SC, Gersh BJ, Brown RD Jr, Rosales AG, Munger TM, Shen WK, Hammill SC, Friedman PA. The natural history of lone atrial flutter. Ann Intern Med. 2004 Feb 17;140(4):265-8. doi: 10.7326/0003-4819-140-4-200402170-00008. PMID 14970149
- [Background] Bun SS, Latcu DG, Marchlinski F, Saoudi N. Atrial flutter: more than just one of a kind. Eur Heart J. 2015 Sep 14;36(35):2356-63. doi: 10.1093/eurheartj/ehv118. Epub 2015 Apr 2. PMID 25838435
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Sehar N, Mears J, Bisco S, Patel S, Lachman N, Asirvatham SJ. Anatomic guidance for ablation: atrial flutter, fibrillation, and outflow tract ventricular tachycardia. Indian Pacing Electrophysiol J. 2010 Aug 10;10(8):339-56. PMID 20811537
- [Background] Da Costa A, Faure E, Thevenin J, Messier M, Bernard S, Abdel K, Robin C, Romeyer C, Isaaz K. Effect of isthmus anatomy and ablation catheter on radiofrequency catheter ablation of the cavotricuspid isthmus. Circulation. 2004 Aug 31;110(9):1030-5. doi: 10.1161/01.CIR.0000139845.40818.75. Epub 2004 Aug 23. PMID 15326078
- [Background] Schernthaner C, Haidinger B, Brandt MC, Kraus J, Danmayr F, Hoppe UC, Strohmer B. The influence of cavotricuspid isthmus length on total radiofrequency energy to cure right atrial flutter. Kardiol Pol. 2016;74(3):237-43. doi: 10.5603/KP.a2015.0159. Epub 2015 Aug 25. PMID 26305365
- [Background] Cohen TJ, Ibrahim B, Lazar J, Rosen J, Klein J. Utility of intracardiac echocardiography (ICE) in electrophysiology: ICEing the CAKE (catheter ablation knowledge enhancement). J Invasive Cardiol. 1999 Jun;11(6):364-8. PMID 10745552